CLINICAL TRIAL: NCT00638859
Title: Evaluation of the Safety, Pharmacokinetics, Efficacy, and Acceptability of HMR3647 20 mg/kg qd for 5-7 Days With Community-Acquired Pneumonia (CAP) in Children (Multicenter, Open Label, Noncomparative Study)
Brief Title: Japanese Study Evaluating the Effects of Telithromycin in Children With Community-Acquired Pneumonia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EFC6369; HMR3647B/3101
Record Dates: First submitted 2008-03-12; First posted 2008-03-19 (Estimated); Last update posted 2009-10-02 (Estimated); Status verified 2009-10

CONDITIONS: Pneumonia
Keywords: Community-Acquired pneumonia; CAP; children; Child
MeSH Terms: conditions — Pneumonia; Community-Acquired Pneumonia | interventions — telithromycin

INTERVENTIONS:
Drug: Telithromycin (HMR3647)

SUMMARY:
The primary objective is to assess the safety of telithromycin (HMR3647) 20 mg/kg qd for 5-7 days in children with community-acquired pneumonia (CAP).

Secondary objectives are to assess Pharmacokinetics, Efficacy and Acceptability of telithromycin 20 mg/kg qd for 5-7 days in children with CAP.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are weighing 40 kg or less. If female, premenarchal status is required.
* Subjects who are diagnosed with CAP based on chest X-ray showing the presence of a new infiltrate, clinical symptoms, and laboratory findings.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 6 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2004-03; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Safety evaluation: presence/absence of subjective/objective symptoms and abnormal laboratory findings

SECONDARY OUTCOMES:
Clinical efficacy: change in the symptoms and signs
Acceptability: compliance and willingness to take medication
Pharmacokinetics: plasma concentrations of telithromycin

CONTACTS AND LOCATIONS:
Overall Officials: CSD, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Tokyo, Japan